CLINICAL TRIAL: NCT04691999
Title: EFFECT-BC: The EFFECT of Intermittent Fasting on Body Composition in Women With Breast Cancer
Brief Title: The Effect of Intermittent Fasting on Body Composition in Women With Breast Cancer
Acronym: EFFECT-BC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is leaving Duke for a position in another state.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00107216
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: intermittent fasting
MeSH Terms: conditions — Breast Neoplasms; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent Fasting (Experimental): All participants will either delay their first meal of the day or advance their last meal to achieve an approximate 16-18 hour fasting period four times per week.
  Interventions: Behavioral: Intermittent Fasting

INTERVENTIONS:
Behavioral: Intermittent Fasting — 16-18 hour fasting period four times per week

SUMMARY:
The objective of this study is to evaluate intermittent fasting after the treatment of breast cancer with surgery and radiation therapy. All participants will either delay their first meal of the day or advance their last meal to achieve an approximate 16-18 hour fasting period four times per week. Over six months, the innovative protocol will 1) assess adherence, and is expected to 2) improve body composition, quality of life and inflammatory and metabolic variables linked with outcomes after breast cancer treatment. The long-term goal of this project is to incorporate this dietary strategy as a standard component of care for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast stage I-III
* completed any chemotherapy prior to initiation of the trial (adjuvant endocrine therapy is permitted)
* BMI > 25 kg/m2 or body fat% greater or equal to 31%
* have a schedule amenable to nutrition and dietitian counseling described within the study protocol as determined by the treating radiation oncologist
* have access to the internet and email with capability to join Zoom calls

Exclusion Criteria:

* Metastatic breast cancer
* Currently receiving chemotherapy
* Uncontrolled hypertension or diabetes, defined as systolic blood pressure over 149, diastolic blood pressure over 99, or hemoglobin A1c greater than 8.9.
* Diabetic condition requiring the usage of insulin

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is not based on self-representation of gender identity
Enrollment: 0 (Actual)
Dates: Start 2021-12-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to the intermittent fasting program | 6 months
  as determined by the proportion of fasting days met divided by the total fasting days planned for each participant
Change in body fat | baseline, 6 months
  as measured by mean change in percent body fat between baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD CSCS, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No